CLINICAL TRIAL: NCT02697617
Title: Use of Low Dose Pioglitazone to Treat Autosomal Dominant Polycystic Kidney
Brief Title: Use of Low Dose Pioglitazone to Treat Autosomal Dominant Polycystic Kidney Disease
Acronym: PIOPKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Sharon Moe, MD, Stuart A. Kleit Professor of Medicine, Director, Division of Nephrology, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IndianaU 1308084213; FD-R-004826-01-A2 (Other: FDA Orphan Products Development Ad Hoc Panel Review)
Record Dates: First submitted 2015-10-30; First posted 2016-03-03 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): Subject will be on placebo
  Interventions: Drug: Placebo
- Pioglitazone Arm (Active Comparator): Subject will be on pioglitazone
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone
  Other Names: Actos
  Arms: Pioglitazone Arm
Drug: Placebo — Placebo
  Arms: Placebo Arm

SUMMARY:
Funding Source - FDA OOPD

Pioglitazone is currently used in clinical practice to treat diabetes and this study will examine the potential use of a low dose of the same drug for the treatment of polycystic kidney disease. The purpose of this study is to determine whether the diabetes drug pioglitazone (Actos) is a safe and effective treatment of autosomal dominant polycystic kidney disease when treated in its early stages. Pioglitazone is approved by the FDA for the treatment of diabetes. Pre-clinical models of polycystic kidney disease have shown that low dose treatment with pioglitazone decreases the growth of the cysts. The studies also suggest that effective pioglitazone dosing for polycystic kidney disease may be lower than that used to treat diabetes. The purpose of this study is to see if pioglitazone might slow cyst disease in humans.

DETAILED DESCRIPTION:
Patients will be randomize to placebo or 15 mg pioglitazone for 12 months, and then be crossed over to the other arm. Patients will undergo MRI of the liver and kidney and MRspectroscopy of the lumbar spine (if they choose as this is ancillary study) three times during the study. Assessments will be every 3 months and include blood work, blood pressure, and body water assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with autosomal dominant polycystic kidney disease (ADPKD) aged 18-55
* estimate glomerular filtration rate (GFR) at or above ≥ 50 ml/min/1.73 m2 by any GFR formula
* Normal liver enzymes (ALT/AST)
* fasting blood glucose between 70 and120
* for female patients, a willingness to use double contraception to avoid pregnancy while in study
* able to give informed consent
* In the opinion of the investigator, high likelihood of progressive kidney disease

Exclusion Criteria:

* diabetes, defined as any of the following: fasting blood sugar > 130 times two, HgbA1C > 7, on any blood sugar lowering medication, or past diagnosis of diabetes not occurring during pregnancy
* uncontrolled hypertension as determined by the examining physician
* history of impaired systolic function (ejection fraction < 50%) by previous echocardiogram or known ischemic cardiovascular disease
* findings suggestive of a kidney disease other than ADPKD
* systemic illness requiring immunosuppressive or anti-inflammatory agents
* congenital absence of a kidney or history of a total nephrectomy
* history of cyst reduction or partial nephrectomy
* history of renal cyst aspiration within the previous year
* History of bladder cancer, or gross hematuria
* inability to undergo MRI due to implantable devices or foreign objects that preclude MRI
* active renal transplant
* allergy or sensitivity to any of the components of the test materials
* institutionalized
* currently pregnant or plans to become pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Moe, 317-944-7580, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Age 18-55 years old, with known autosomal dominant polycystic kidney disease (ADPKD), estimated glomerular filtration rate (eGFR) > 50 ml/min/m2 on recent labs, and no history of diabetes were identified using international disease codes (ICD-9) code for cystic kidney disease by search of electronic medical records or through advertisements and letters sent to Nephrologists.
Pre-assignment Details: Patients who fulfilled the initial screening underwent further screening with a baseline magnetic resonance imaging (MRI) and randomized to pioglitazone or placebo providing the total kidney volume (TKV) was ≥675 ml (18-25 years old), ≥ 900 ml (26-35 years old), and ≥ 1350 ml (36-55 years old).
Groups:
- PIO Then PLACEBO: Sequence Pioglitazone then Placebo
- Placebo Then PIO: sequence placebo then pioglitazone
Period: Overall Study
Arm/Group | PIO Then PLACEBO | Placebo Then PIO
Started | 9 | 9
Completed | 8 (15 completed both arms) | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: 18 patients randomized to either pioglitazone for 12 months and then placebo for 12 months and then cross over to the other arm. So baseline data represents both arms
Groups:
- All Study Participants: at randomization to sequence 1 (pioglitazone 15 mg) or placebo for cross over study
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 18
estimated glomerular filtration rate (eGFR) by CKD-epi [Mean (Standard Deviation); unit: ml/min/m2] | 86 (27)
right kidney volume [Mean (Standard Deviation); unit: ml] | 965 (636)
left kidney volume [Mean (Standard Deviation); unit: ml] | 1078 (652)

OUTCOME MEASURES:

1. Primary Outcome: Safety: Total Body Water
Description: Bioimpedance analysis (BIA)(Ohms); Increase in BIA in Ohms indicates a decrease in total body water
Time Frame: average of 4 measures in each 12 month arm
Population: All patients randomized
Measure: Mean (95% Confidence Interval); unit: Ohms
Groups:
- Pioglitazone; Placebo: Total body water
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 18 | 18
Ohms | 45.78 [39.19 to 52.36] | 44.17 [37.96 to 50.39]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority; p = 0.024, Paired t-test — First analyzed using a Linear Mixed Model to assess if there were carryover effects and then subsequently analyzed using paired t-tests to compare the mean differences between treatments

2. Primary Outcome: Efficacy: Percent Change in Total Kidney Volume
Description: Change in total kidney volume by Magnetic Resonance Imaging (MRI) from beginning to end of the 12 months
Time Frame: Baseline, end of year 1, and end of year 2
Population: Those who completed both arms
Measure: Mean (95% Confidence Interval); unit: percentage of change
Groups:
- Pioglitazone 15 mg Daily: Patients who completed both arms, data from the 12 months of pioglitazone treatment
- Placebo po Daily: of patients who finished both arms, the results from the placebo arm
Arm/Group | Pioglitazone 15 mg Daily | Placebo po Daily
Number analyzed (Participants) | 15 | 15
percentage of change | 4.35 [0.84 to 7.86] | 7.85 [3.6 to 12.11]
Statistical Analysis 1: Comparison: Pioglitazone 15 mg Daily vs Placebo po Daily; Test type: Superiority; p = 0.14, Paired t-test — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Safety: Hypoglycemia
Description: number of patients with blood sugar < 70 mg/dl
Time Frame: measured quarterly for 12 months in pioglitazone and same in placebo
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Groups:
- Pioglitazone 15 mg: All patients taking pioglitazone
- Placebo: all patients taking placebo
Arm/Group | Pioglitazone 15 mg | Placebo
Number analyzed (Participants) | 18 | 18
Participants | 1 | 1

4. Secondary Outcome: Safety: Elevated Liver Function Tests
Description: Number of patients with elevated liver test (ALT or AST) > 2 times upper limit of normal
Time Frame: measured quarterly over 12 months for each arm
Population: All patients who were randomized, regardless of whether they completed both arms
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone 15 mg | Placebo
Number analyzed (Participants) | 18 | 18
Participants | 0 | 1
Statistical Analysis 1: Comparison: Pioglitazone 15 mg vs Placebo; Test type: Other; comparison by paired t-test

5. Secondary Outcome: Efficacy: Glomerular Filtration Rate
Description: average estimated glomerular filtration rate by chronic kidney disease (CKD) epidemiologic (epi) formula measured quarterly
Time Frame: average of 4 values over 12 months
Population: All patients that completed both arms.
Measure: Mean (95% Confidence Interval); unit: ml/min/m2
Arm/Group | Pioglitazone 15 mg | Placebo
Number analyzed (Participants) | 15 | 15
ml/min/m2 | 75.5 [62 to 89] | 78.1 [64 to 92]
Statistical Analysis 1: Comparison: Pioglitazone 15 mg vs Placebo; Test type: Superiority; p = 0.15, Paired t-test — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Efficacy Blood Pressure
Description: mean systolic and diastolic blood pressure
Time Frame: average of 4 measures over 12 months
Population: All patients that completed both arms
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Pioglitazone 15 mg | Placebo
Number analyzed (Participants) | 15 | 15
mmHg
  systolic blood pressure | 127 [124 to 130] | 129 [124 to 134]
  diastolic blood pressure | 83 [81 to 86] | 82 [82 to 89]
Statistical Analysis 1: Comparison: Pioglitazone 15 mg vs Placebo; Test type: Superiority; p = 0.4, paired t test — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Bone Marrow Fat
Description: We will assess change in bone marrow fat by MR spectroscopy as an ancillary study to be done at the same time as MRI; will not be done due to person leaving institution.
Time Frame: Baseline, end of year 1, and end of year 2
Population: The MRIs were done, but could not be analyzed as requires special expertise and software.
Arm/Group | Pioglitazone 15 mg Daily | Placebo po Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Pioglitazone: 15 mg po daily
- Placebo: Over encapsulated (identical appearing) placebo
Arm/Group | Pioglitazone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 3/18
Other Adverse Events (participants affected / at risk) | 13/18 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=18) | Placebo (N=18)
hospitalization (Hepatobiliary disorders) | 0 (0) | 1 (1) — pancreatitis
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
surgery (Gastrointestinal disorders) | 0 (0) | 1 (1) — elective surgery/gastric banding
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=18) | Placebo (N=18)
headache (Nervous system disorders) | 8 (12) | 9 (11)
dizziness (Nervous system disorders) | 4 (6) | 3 (6)
infection (Infections and infestations) | 13 (38) | 15 (30)
gastrointestinal symptom (Gastrointestinal disorders) | 6 (9) | 5 (10)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (17) | 9 (23)
urinary tract infection or pain (General disorders) | 7 (12) | 9 (18) — or cyst rupture

LIMITATIONS AND CAVEATS:
The major limitation is the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT02697617/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02697617/Prot_SAP_001.pdf